CLINICAL TRIAL: NCT01706133
Title: Elderly in Emergency Services: Effectiveness of an Intervention to Improve Health Outcomes
Brief Title: An Intervention for Elderly in Emergency Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Maria del Carmen Garcia-Pena, Head, Research Unit on Aging, Coordinación de Investigación en Salud, Mexico
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: R-201 l-785-056
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Stroke; Ischemic Attack; Diabetes Mellitus; Hypertension; Fragility
Keywords: Frailty, emergency services, elderly
MeSH Terms: conditions — Stroke; Diabetes Mellitus; Hypertension; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Basal phase (No Intervention): Integrated measurement of all variables involved impact and frequency of prior use of health services and specifically to the emergency room, service access, patient characteristics, features for the classification of frailty, cognitive impairment and depression, why consultation, triage scale level on admission to the service and to the service variables in terms of length of stay, diagnosis and medical management, and related services with internal consultants percentage of inpatients discharged or deceased, in further analysis the researchers undertake group estimating frequency of use and the identification of factors associated with the use of emergency departments and adverse events
  Interventions: Other: Factors associated with the use of emergency departments

INTERVENTIONS:
Other: Factors associated with the use of emergency departments — Participants who were assigned to the intervention will be evaluated jointly by the medical service by a medical specialist in geriatrics and a nurse trained in gerontology and geriatrics. The doctor will monitor the apparition and / or aggravation of any geriatric syndromes already established by the specialty in geriatrics, namely, polypharmacy, delirium, dementia, depression, risk of falls, etc.. The nurse will monitor and follow up in four areas I. medical issues (pressure ulcers, infusion, mobility); II. Mental and emotional state and coping strategies with hospitalization; III. functionality, and IV. Atmosphere (A. Service status, architectural difficulties for mobility, bathing etc. B. Support Network, caregiver, and C. hardship)

SUMMARY:
-Can a scheme based on inter geriatricians visiting nurse consultants and reduce negative impacts on the health of elderly over 70 years ?

DETAILED DESCRIPTION:
- Usual care as the comparison group

Usual care or standard refers to those processes or services that the elderly claimant receives the IMSS services network, after the acute phase of their illness has been stabilized and is defined that can be discharged from the emergency department, following clinical and therapeutic recommendations for improving their health.

* Elders risk population for emergency

The aging population brings a major change in health conditions and social conditions around the elderly, the analysis of the elderly population is considered according to functionality and risks of old age, when it comes to care services emergency, care becomes more critical as the elderly are older, have been identified adults of 70 and over as more vulnerable to health services, especially for the emergency services as they do not exhibit classic patterns to acute events of prevalent diseases.

* Functionality and dependence

The commitment of the functionality in adults older than 65 may be present in 5% of cases, while in over 70 years this figure rises to 50% or more. Functional impairment may be a "marker" of the effect of systemic disease on the patient and is also an indicator of severity of disease because it measures the ability of independence

The accumulation of normal aging characteristics define a threshold, which once pierced, tends to increase the propensity for loss of functional abilities due to aging. However, not everyone ages the same way, since factors such as inherited genetic capital, especially the accumulation of risks associated with lifestyle and work activities, and the opportunity to identify the disease in its period latency coupled with the accessibility and use of health services, can delay or exacerbate the loss of functionality and increase the dependency of the elderly.

* Quality of life of older

Frailty in the elderly is a state of increased susceptibility due to less booking multiple physiological systems resulting in lower resilience, negative energy balance, sarcopenia, decreased strength and reduced exercise tolerance. Frailty is associated with adverse health outcomes such as institutionalization, falls, reduced performance status and increased mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults 70 and over.
* Both sexes
* Affiliation force in the IMSS
* Attending spontaneously or referred to the emergency department of hospitals in the study.
* Agree to participate in the study phase in observational or intervention by signed written informed consent

Exclusion Criteria:

1. Adults 70 and older whose income is service by:

   a. A very serious acute condition with imminent risk to life and requires immediate emergency care, cataloged by the Triage system marked by the IMSS as Red or (state the patient's functional impairment characterized by high and low, with imminent risk life or the integrity and function of some of their organs and requires immediate medical attention since his arrival to the emergency room) or require emergency care (patient condition characterized by acute and severe functional impairment, life-threatening or the integrity and function of some of their organs and requires medical attention within the next 10 minutes after arrival at the emergency department).
   * An automobile accident
   * Burn-grade II or III
   * Partial or total unconsciousness
   * Severe cognitive impairment
2. Individuals who do not agree to participate in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in hand grip strength (HS) as a physical performance test | Basal and Six months
  A standardized technique and digital dynamometers (Exacta TM) wil lbe used, and the best result of two tests in the dominant hand will be used for analysis. No cut-off points will be applied; instead the variable will be assessed as a continuous one with kilograms as the units of measure.

SECONDARY OUTCOMES:
Evaluation of individual and institutional impact | Six Months
  Evaluate the impact of a scheme based on internal consultation geriatricians and home visiting nurses oriented elders 70 and over, in terms of individual outcomes and health services:
  a. Individual Impacts:
  a.1 Primary:
  • Fragility

OTHER OUTCOMES:
Quantify hospital readmissions | One Year
  Estimate the readmission to hospital adverse events in adults older than 70 years, underwent surgery and its comparison group from discharge from service

CONTACTS AND LOCATIONS:
Overall Officials: Carmen García-Peña, PhD, Principal Investigator — Epidemiological Research Unit and Health Services. XXI Century National Medical Center; Sergio Sánchez García, PhD, Study Chair — Epidemiological Research Unit and Health Services. XXI Century National Medical Center; Teresa Juarez Cedillo, PhD, Study Chair — Epidemiological Research Unit and Health Services. XXI Century National Medical Center; Rogelio Moncada Tobias, Doctor, Study Chair — Emergency Service. General Hospital Zone No.2; Nubia Franco Alvarez, Doctor, Study Chair — Internal Medicine. General Hospital Zone No. 2; José García González, Master, Study Chair — Department of Nephrology. Regional General Hospital No. 1; Ulises Pérez Zepeda, Master, Study Chair — Institute of Geriatrics; Leslie Viridiana Robles Jiménez, Doctor, Study Chair — National Institute of Psychiatry
Locations (1):
- XXI Century National Medical, Mexico City, Mexico City, Mexico